CLINICAL TRIAL: NCT05104333
Title: A Post-marketing Clinical Study of a Third Dose of the Inactivated SARS-CoV-2 Vaccine (Vero Cells) (Produced in Beijing): Immunogenicity, Safety and Antibody Persistence Assessments in Patients With Hypertension and/or Diabetes
Brief Title: Evaluation of Immunogenicity, Safety and Antibody Persistence of COVID-19 Booster Vaccine (Produced in Beijing) in Patients With Hypertension and/or Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Guizhou Center for Disease Control and Prevention (Other); Hunan Provincial Center for Disease Control and Prevention (Other); Center for Disease Control and Prevention, Fujian (Other); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COVAX BOOSTER (HT/DM)-Beijing
Record Dates: First submitted 2021-10-30; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Serum testing technicians will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0-1-4 schedule group (Experimental): Subjects receive the booster vaccine 3 months after the second dose.
  Interventions: Biological: Covid-19 vaccine (0-1-4 schedule)
- 0-1-6 schedule group (Experimental): Subjects receive the booster vaccine 5 months after the second dose.
  Interventions: Biological: Covid-19 vaccine (0-1-6 schedule)

INTERVENTIONS:
Biological: Covid-19 vaccine (0-1-4 schedule) — Subjects receive the booster vaccine 3 months after the second dose.
  Arms: 0-1-4 schedule group
Biological: Covid-19 vaccine (0-1-6 schedule) — Subjects receive the booster vaccine 5 months after the second dose.
  Arms: 0-1-6 schedule group

SUMMARY:
To evaluate the post-marketing immunogenicity, safety and antibody persistence of the third dose (booster) of Covid-19 vaccine in patients aged 60 years or older with hypertension and/or diabetes.

DETAILED DESCRIPTION:
After giving informed consent, patients with hypertension, patients with diabetes, patients with both diseases, and healthy controls, all aged 60 years or older, are given a third doses of the inactivated SARS-CoV-2 vaccine (Vero cells).

These subjects are all from the "COVAX (HT/DM)-Beijing" clinical trial (NCT05065879). 50% of them receive the booster vaccine 3 months after the second dose (0-1-4 schedule); 50% of them receive the booster vaccine 5 months after the second dose (0-1-6 schedule).

Venous blood samples are collected before the booster dose and on day 28 after the booster dose to evaluate the immunogenicity of the vaccine.

Venous blood samples are also collected on day 84/168/252/336 after the booster dose to evaluate the antibody persistence of the vaccine.

Adverse events are actively recorded on a diary card once daily from day 0 to day 7 and once from day 8 to day 21 after the booster dose. Serious adverse events (SAE) are collected within 6 months after the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Participate in the clinical trial "NCT05065879".
* ≥60 years old individuals with full civil capacity.
* Clinically confirmed body temperature of <37.3°C before enrolling in this study.
* Able and willing to participate in the study plan during the entire study and follow-up period.
* Capable of understanding the study procedures, willing to sign the informed consent form, and able to comply with the requirements of the clinical study protocol.
* Inclusion criteria for patients with hypertension and/or diabetes: Hypertension and/or diabetes definitively diagnosed by a community-level or higher medical institution. Patients with hypertension: systolic pressure <160 mmHg and diastolic pressure <100 mmHg on the day of immunization achieved by lifestyle adjustment and/or drug treatment; patients with diabetes: fasting glucose ≤13.9 mmol/L on the day of (or within 3 days before) immunization achieved by lifestyle adjustment and/or drug treatment

Exclusion Criteria:

* Previously confirmed or asymptomatic COVID-19 patient.
* Has been immunized with a SARS-CoV-2 vaccine.
* Illiterate.
* Known allergy to any ingredient (including excipient) of this product.
* Received non-specific immunoglobulin injection within 1 month before enrollment.
* Received a live attenuated vaccine within 1 month before immunization or other vaccine within 14 days before immunization.
* Previous serious allergy to vaccine (e.g., acute allergic reaction, urticaria, angioedema, and dyspnea).
* Has uncontrolled epilepsy and other progressive neurological disorders; history of Guillain-Barré syndrome.
* Severe respiratory disorders, severe hepatic and renal diseases, malignancies, and various acute diseases or acute onset of chronic diseases.
* Diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases.
* Definitively diagnosed with thrombocytopenia or history of other coagulation disorders that may cause subcutaneous injection to be contraindicated.
* Currently experiencing acute complications (ketoacidosis, hyperosmolar state, lactic acidosis, etc.) of diabetes; or within 2 weeks after recovery from these complications.
* Other physical conditions judged by the investigator that render the patient unsuitable for participation in the clinical study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | Up to 28 days after the booster dose
  the rate of positive seroconversion against coronavirus
Neutralizing antibody level | Up to 28 days after the booster dose
  neutralizing antibody level against coronavirus
Neutralizing antibody level | Up to 84 days after the booster dose
  neutralizing antibody level against coronavirus
Neutralizing antibody level | Up to 168 days after the booster dose
  neutralizing antibody level against coronavirus
Neutralizing antibody level | Up to 252 days after the booster dose
  neutralizing antibody level against coronavirus
Neutralizing antibody level | Up to 336 days after the booster dose
  neutralizing antibody level against coronavirus

SECONDARY OUTCOMES:
Adverse events following vaccination | Up to 6 months after the booster dose
  analyse the incidence of adverse events following immunization, both solicited and unsolicited

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Nan'an Center for Disease Control and Prevention, Quanzhou, Fujian
  - Yong'an Center for Disease Control and Prevention, Sanming, Fujian
  - Youxi Center for Disease Control and Prevention, Sanming, Fujian
  - Songtao Miao Autonomous County Center for Disease Control and Prevention, Tongren, Guizhou
  - Linli County Center for Disease Control and Prevention, Changde, Hunan

IPD SHARING:
Plan to Share IPD: No